CLINICAL TRIAL: NCT01131078
Title: A Randomized, Open-label Study Comparing the Effect of 3 Chemotherapy Regimens Containing Avastin on Time to Disease Progression in Patients With Metastatic Colorectal Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination Chemotherapy in Patients With Metastatic Cancer of the Colon or Rectum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18524
Record Dates: First submitted 2010-04-20; First posted 2010-05-26 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Irinotecan

ARMS (3):
- Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) (Experimental): Bevacizumab was administered as a 7.5 mg/kg intravenous infusion over 30 to 90 minutes on Day 1 of each 3 week cycle. Irinotecan was administered as a 240 mg/m^2 intravenous infusion over 60 minutes (Day 1) every 3 weeks. Capecitabine was administered orally at a dose of 1000 mg/m^2 twice daily (Day 2 to 15). Cycle length was 3 weeks consisting of 2 weeks of capecitabine treatment followed by 1 week without treatment up to 6 cycles. After 6 cycles, participants with objective response or SD were treated with bevacizumab alone until unacceptable toxicity, PD, or participant withdrawal.
  Interventions: Drug: Bevacizumab [Avastin]; Drug: Capecitabine; Drug: Irinotecan
- Bevacizumab + Capecitabine (1250 mg/m^2) (Experimental): Bevacizumab was administered as a 7.5 mg/kg intravenous infusion over 30 to 90 minutes on Day 1 of each 3 week cycle in combination with capecitabine administered orally at 1250 mg/m^2 twice daily (Day 1 to 14). Cycle length was 3 weeks with 2 weeks of capecitabine treatment followed by 1 week without treatment up to 6 cycles. After 6 cycles, participants with objective response or SD were treated with bevacizumab alone until unacceptable toxicity, PD, or participant withdrawal.
  Interventions: Drug: Bevacizumab [Avastin]; Drug: Capecitabine
- Bevacizumab + Capecitabine (650 mg/m^2) (Experimental): Bevacizumab was administered as a 7.5 mg/kg intravenous infusion over 30 to 90 minutes on Day 1 of each 3 Week cycle in combination with capecitabine administered orally at 650 mg/m^2 twice daily (Day 1 to 21). Cycle length was 3 weeks with 3 weeks of capecitabine treatment without interruptions. Participants received the same regimen until unacceptable toxicity, PD, or participant withdrawal.
  Interventions: Drug: Bevacizumab [Avastin]; Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab [Avastin] — Bevacizumab was administered as a 7.5 mg/kg intravenous infusion over 30 to 90 minutes on Day 1 of each 3 week cycle.
  Other Names: Avastin
Drug: Capecitabine — Capecitabine was administered orally at a doses of 1000 or 1250, mg/m^2 twice daily (Day 2 to 15) or as 650 mg/m^2 twice daily on Days 1 to 21.
Drug: Irinotecan — Irinotecan was administered as a 240 mg/m^2 intravenous infusion over 60 minutes (Day 1) every 3 weeks.
  Arms: Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2)

SUMMARY:
A study of Avastin (bevacizumab) in combination chemotherapy in patients with metastatic cancer of the colon or rectum. The anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* colon or rectal cancer, with metastases;
* >=1 measurable lesion.

Exclusion Criteria:

* previous systemic treatment for advanced disease;
* radiotherapy to any site within 4 weeks before study;
* daily aspirin (>325 mg/day), anticoagulants, or other medications known to predispose to gastrointestinal ulceration;
* co-existing malignancies or malignancies diagnosed within last 5 years (except basal cell cancer or cervical cancer in situ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2005-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (40):
- Italy (40):
  - Paola, Calabria
  - Benevento, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Carpi, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Latisana, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Latina, Lazio
  - Rome, Lazio
  - Brescia, Lombardy
  - Busto Arsizio, Lombardy
  - Casalpusterlengo, Lombardy
  - Cremona, Lombardy
  - Gorgonzola, Lombardy
  - Lecco, Lombardy
  - Legnago, Lombardy
  - Mantova, Lombardy
  - Milan, Lombardy
  - Pavia, Lombardy
  - Saronno, Lombardy
  - Sondrio, Lombardy
  - Treviglio, Lombardy
  - Varese, Lombardy
  - Novara, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Catania, Sicily
  - Palermo, Sicily
  - Ancona, The Marches
  - Bolzano, Trentino-Alto Adige
  - Florence, Tuscany
  - Grosseto, Tuscany
  - Pisa, Tuscany
  - Prato, Tuscany
  - Terni, Umbria
  - Camposampiero, Veneto
  - Este, Veneto
  - Montecchio Maggiore, Veneto
  - Negrar, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2): Bevacizumab was administered as a 7.5 milligrams per kilogram (mg/kg) intravenous infusion over 30 to 90 minutes on Day 1 of each 3 week cycle. Irinotecan was administered as a 240 milligrams per meter squared (mg/m^2) intravenous infusion over 60 minutes (Day 1) every 3 weeks. Capecitabine was administered orally at a dose of 1000 mg/m^2 twice daily (Day 2 to 15). Cycle length was 3 weeks consisting of 2 weeks of capecitabine treatment followed by 1 week without treatment up to 6 cycles. After 6 cycles, participants with objective response or stable disease (SD) were treated with bevacizumab alone until unacceptable toxicity, progressive disease (PD), or participant withdrawal.
Period: Overall Study
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Started | 101 | 102 | 103
Completed | 0 | 1 | 1
Not Completed | 101 | 101 | 102
Not completed — Adverse Event | 22 | 12 | 17
Not completed — Progressive Disease | 58 | 77 | 71
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 3
Not completed — Non-compliance | 3 | 0 | 0
Not completed — Physician Decision | 10 | 6 | 8
Not completed — Death | 4 | 0 | 2
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants were included in the Intent-to-Treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2) | Total
Number analyzed (Participants) | 101 | 102 | 103 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.60 (9.35) | 61.46 (10.22) | 61.01 (10.10) | 61.36 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 63 | 174
  Male | 43 | 49 | 40 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression or Death
Description: Disease progression was defined according to National Cancer Institute (NCI) guidelines and best clinical practices.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population;
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab + Capecitabine (1250 mg/m^2): Bevacizumab was administered as a 7.5 mg/kg intravenous infusion over 30 to 90 minutes on Day 1 of each 3-week cycle in combination with capecitabine administered orally at 1250 mg/m^2 twice daily (Day 1 to 14). Cycle length was 3 weeks with 2 weeks of capecitabine treatment followed by 1 week without treatment up to 6 cycles. After 6 cycles, participants with objective response or SD were treated with bevacizumab alone until unacceptable toxicity, PD, or participant withdrawal.
- Bevacizumab + Capecitabine (650 mg/m^2): Bevacizumab was administered as a 7.5 mg/kg intravenous infusion over 30 to 90 minutes on Day 1 of each 3-week cycle in combination with capecitabine administered orally at 650 mg/m^2 twice daily (Day 1 to 21). Cycle length was 3 weeks with 3 weeks of continuous capecitabine treatment. Participants received the same regimen until unacceptable toxicity, PD, or participant withdrawal.
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 101 | 102 | 103
percentage of participants | 86.14 | 90.20 | 88.35

2. Secondary Outcome: Percentage of Participants Who Died
Description: Overall survival is defined as the time from date of randomization until death from any cause
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 101 | 102 | 103
percentage of participants | 67.33 | 71.57 | 73.79

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of randomization until death from any cause; Kaplan-Meier estimates were used for analysis.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; Only participants with an event (death) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 68 | 73 | 76
months | 22.75 [18.94 to 26.63] | 19.76 [18.38 to 24.00] | 18.02 [14.76 to 20.61]

4. Secondary Outcome: Percentage of Participants With Treatment Failure
Description: Treatment failure is defined as discontinuation of treatment for any reason, including disease progression, death, treatment toxicity, insufficient therapeutic response, failure to return, refusing treatment, being unwilling to cooperate and withdrawing consent.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 101 | 102 | 103
percentage of participants | 100.0 | 99.02 | 99.03

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as a composite endpoint measuring time from date of randomization to discontinuation of treatment for any reason, including disease progression, death, treatment toxicity, insufficient therapeutic response, failure to return, refusing treatment, being unwilling to cooperate and withdrawing consent. Analysis was performed using Kaplan-Meier estimates.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; only participants with a treatment failure event were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 101 | 101 | 102
months | 6.67 [5.82 to 7.56] | 6.87 [5.49 to 8.38] | 5.75 [4.34 to 7.27]

6. Secondary Outcome: Percentage of Participants With Progression Excluding Deaths
Description: The failure event was defined as tumor progression excluding deaths due to any reason.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 101 | 102 | 103
percentage of participants | 71.29 | 81.37 | 75.73

7. Secondary Outcome: Time to Progression Excluding Deaths
Description: The failure event was defined as tumor progression excluding deaths due to any reason. Kaplan-Meier estimates were used for analysis.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; Only participants with a time to progression event (excluding deaths) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 72 | 83 | 78
months | 8.81 [7.66 to 10.82] | 8.48 [6.90 to 8.84] | 7.40 [4.87 to 9.17]

8. Secondary Outcome: Percentage of Participants With Progression Excluding Deaths Not Related to Underlying Cancer
Description: The failure event was defined as tumor progression excluding only deaths not related to underlying cancer.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 101 | 102 | 103
percentage of participants | 81.19 | 90.20 | 85.44

9. Secondary Outcome: Time to Progression Excluding Deaths Not Related to Underlying Cancer
Description: The failure event was defined as tumor progression excluding only deaths not related to underlying cancer. Kaplan-Meier estimates were used for analysis.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; only participants with a time to progression event (excluding deaths not related to underlying cancer) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 82 | 92 | 88
months | 8.68 [7.59 to 9.90] | 8.32 [6.74 to 8.75] | 7.27 [4.57 to 9.11]

10. Primary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from date of randomization until objective tumor progression or death due to any cause. It includes deaths and thus can be correlated to overall survival.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; only those participants with an event of disease progression or death were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 87 | 92 | 91
months | 8.35 [7.23 to 9.60] | 8.15 [6.74 to 8.75] | 7.27 [4.57 to 8.98]

11. Secondary Outcome: Percentage of Participants by Best Overall Response
Description: Best overall response is defined as the best response recorded from the date of randomization until disease progression or recurrence. Complete response (CR): at least 2 determinations of CR at least 4 weeks apart before progression; Partial response (PR): at least 2 determinations of PR at least 4 weeks apart before progression; Stable disease (SD): at least one SD assessment; Progressive Disease (PD): Disease progression or death due to underlying cancer. CR: Complete disappearance of all target lesions; PR: At least 30% decrease in the sum of the longest diameter of all target lesions taking as reference the baseline sum of all target lesions; PD: At least 20% decrease in the sum of the longest diameter of all target lesions taking as reference the baseline sum of longest diameter of all target lesions or the appearance of one or more new lesions; SD: Neither sufficient shrinkage to qualify for CR or PR or increase in lesions;
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; All participants with evaluable data were included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 91 | 92 | 94
percentage of participants
  CR | 5.49 | 1.09 | 5.32
  PR | 46.15 | 32.61 | 28.72
  SD | 39.56 | 52.17 | 45.74
  PD | 8.79 | 14.13 | 20.21

12. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR or PR
Description: CR: Complete disappearance of all target lesions; PR: At least 30% decrease in the sum of the longest diameter of all target lesions taking as reference the baseline sum of all target lesions;
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; All participants with evaluable data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 91 | 92 | 94
percentage of participants | 52.0 [41.0 to 62.0] | 34.0 [24.0 to 44.0] | 34.0 [25.0 to 45.0]

13. Secondary Outcome: Percentage of Participants With Stable Disease
Description: Stable disease rate was the proportion of participants who achieved CR, PR, or SD.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; All participants with evaluable data were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 91 | 92 | 94
percentage of participants | 91.0 [83.0 to 96.0] | 86.0 [77.0 to 92.0] | 80.0 [70.0 to 87.0]

14. Secondary Outcome: Percentage of Participants With Progressive Disease Within 12 Weeks From Start of Treatment
Description: Early progression was the proportion of participants with progressive disease within 12 weeks from the start of treatment.
Time Frame: Randomization, Weeks 3, 6 and 9, and 12
Population: ITT Population; All participants with evaluable data were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 91 | 92 | 94
percentage of participants | 9.0 [4.0 to 17.0] | 13.0 [7.0 to 22.0] | 18.0 [11.0 to 27.0]

15. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response included participants who achieved a CR or PR.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; only participants with a best overall response of CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 47 | 31 | 32
months | 6.51 [5.36 to 8.35] | 6.61 [6.15 to 8.28] | 9.12 [6.48 to 16.08]

16. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD was calculated as the number of months the participants remained in CR, PR or SD. Kaplan-Meier estimates were used for analysis.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years or Death
Population: ITT Population; Only participants with a best overall response of CR, PR, or SD were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 83 | 79 | 75
months | 8.81 [7.86 to 10.55] | 8.65 [7.99 to 9.34] | 8.98 [7.30 to 9.99]

17. Secondary Outcome: Duration of Overall Complete Response
Description: Duration of complete response was calculated as the time in months from the date of randomization to the date of first documentation of CR. Kaplan-Meier estimates were used for analysis.
Time Frame: Randomization, Weeks 3, 6 and 9, and every 3 months up to 5 years
Population: ITT Population; Only participants with a best overall response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Number analyzed (Participants) | 5 | 1 | 5
months | 8.35 [5.16 to NA] — Upper limit of the 95% confidence interval was not estimable as the duration of follow-up was not sufficient. | 6.05 [NA to NA] — Number of participants analyzed for this parameter in this treatment group was 1, therefore 95% CI could not be determined. | 12.89 [7.63 to 33.04]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of randomization until the End of Study or until death in safety population. Safety population included all participants who signed informed consent and took at least one dose of each drug of study combination.
Arm/Group | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) | Bevacizumab + Capecitabine (1250 mg/m^2) | Bevacizumab + Capecitabine (650 mg/m^2)
Serious Adverse Events (participants affected / at risk) | 38/100 | 21/99 | 20/102
Other Adverse Events (participants affected / at risk) | 95/100 | 88/99 | 85/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) (N=100) | Bevacizumab + Capecitabine (1250 mg/m^2) (N=99) | Bevacizumab + Capecitabine (650 mg/m^2) (N=102)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 6 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 2
General physical health deterioration (General disorders) | 1 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 1 | 1
Sudden death (General disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Central line infection (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 2 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Device migration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary microemboll (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Toe amputation (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3 | 0
Embolism (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Irinotecan + Capecitabine (1000 mg/m^2) (N=100) | Bevacizumab + Capecitabine (1250 mg/m^2) (N=99) | Bevacizumab + Capecitabine (650 mg/m^2) (N=102)
Anaemia (Blood and lymphatic system disorders) | 18 | 7 | 6
Leukopenia (Blood and lymphatic system disorders) | 7 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 33 | 5 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 2
Conjunctivitis (Eye disorders) | 1 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 21 | 11 | 21
Abdominal pain upper (Gastrointestinal disorders) | 13 | 8 | 8
Constipation (Gastrointestinal disorders) | 12 | 10 | 8
Diarrhoea (Gastrointestinal disorders) | 56 | 34 | 28
Nausea (Gastrointestinal disorders) | 35 | 16 | 26
Stomatitis (Gastrointestinal disorders) | 6 | 10 | 2
Vomiting (Gastrointestinal disorders) | 23 | 13 | 6
Asthenia (General disorders) | 16 | 17 | 20
Fatigue (General disorders) | 14 | 12 | 16
Mucosal inflammation (General disorders) | 13 | 9 | 7
Pyrexia (General disorders) | 30 | 17 | 15
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 | 22 | 26
Alanine aminotransferase increased (Investigations) | 7 | 9 | 12
Aspartate aminotransferase increased (Investigations) | 6 | 8 | 11
Blood alkaline phosphatase increased (Investigations) | 6 | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 9 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4
Headache (Nervous system disorders) | 4 | 7 | 5
Cholinergic syndrome (Nervous system disorders) | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 6 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 2 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 40 | 39
Hypertension (Vascular disorders) | 28 | 29 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 1 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Anal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Ano-rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 4
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 3 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 3 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Oedema peripheral (Gastrointestinal disorders) | 2 | 1 | 1
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Polyp colorectal (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 2
Proctitis (Gastrointestinal disorders) | 2 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 2
Catheter site related reaction (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 3 | 4
Facial pain (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 2
Influenza-like illness (General disorders) | 1 | 3 | 1
Local swelling (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 2 | 1 | 1
Pain (General disorders) | 0 | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 3 | 0 | 2
Abdominal wall infection (Infections and infestations) | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 4 | 1
Dental caries (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 1
Influenza (Infections and infestations) | 3 | 4 | 5
Nail infection (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1
Perianal abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Relapsing fever (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 3 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Intestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood alkaline phosphatase (Investigations) | 1 | 0 | 0
Blood bilirubin (Investigations) | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood creatine increased (Investigations) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 4 | 2
Blood glucose increased (Investigations) | 2 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 2 | 1
Blood sodium increased (Investigations) | 1 | 0 | 0
Coagulation test abnormal (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1
Prothrombin time shortened (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 3 | 0
Weight decreased (Investigations) | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Dysguesia (Nervous system disorders) | 1 | 0 | 1
Migraine without aura (Nervous system disorders) | 2 | 0 | 0
Neuropathy (Nervous system disorders) | 3 | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 3 | 5
Sciatica (Nervous system disorders) | 1 | 3 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 2 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 4 | 4 | 4
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0
Female genital-digestive tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Penis disorder (Reproductive system and breast disorders) | 0 | 3 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 0 | 1
Stent placement (Surgical and medical procedures) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.